CLINICAL TRIAL: NCT05873933
Title: An Investigation of a Multi-Function Skincare Product to Improve Aging, Eczema, and Acne Outcomes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decided to run a different type of research
Sponsor: Hemptress (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20262
Record Dates: First submitted 2023-05-16; First posted 2023-05-24 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Acne; Eczema; Skin Aging
MeSH Terms: conditions — Acne Vulgaris; Eczema

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either one of two groups and their outcomes will be compared separately.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acne and Eczema group (Experimental): Participants who experience regular acne, pimples, eczema, or blemishes. Must use the test products as prescribed. In addition, must be willing to maintain the following skincare routine during the study: (1)Daily cleansing or rinsing of their face in the morning or the evening is sufficient. (2) The option to wear sunscreen if the sunscreen brand is pre-approved - a person who does not wear sunscreen is more desirable. The test product does contain some sun protection (3) Must NOT use any moisturizer besides our oil. Must use the test product in the morning and the evening daily. Must not be using retinoids and must not start using retinoids during the study. Must NOT use oral anti-acne medications/prescriptions.
  Interventions: Other: Hemptress Oil
- Anti-Aging group (Experimental): Participants who experience early-stage wrinkles not treated by topical or oral prescription drugs/medication or over-the-counter products.
  Must use the test products as prescribed. In addition, must be willing to maintain the following skincare routine during the study: (1)Daily cleansing or rinsing of their face in the morning or the evening is sufficient. (2) The option to wear sunscreen if the sunscreen brand is pre-approved - a person who does not wear sunscreen is more desirable. The test product does contain some sun protection (3) Must NOT use any moisturizer besides our oil. Must use the test product in the morning and the evening daily. Must not be using retinoids and must not start using retinoids during the study. Must NOT use oral anti-acne medications/prescriptions.
  Interventions: Other: Hemptress Oil

INTERVENTIONS:
Other: Hemptress Oil — Full ingredient list of the test product: Rubus occidentalis (Black raspberry) seed oil*, Carica papaya (Papaya) seed oil*, Bixa orellana (Annatto) seed oil*, Orbignya oleifera (Babassu) seed oil*, Borago officinalis (Bourrache) seed oil*, Daucus carota (Carrot) seed oil*, Hibiscus sabdariffa (Hibiscus) seed oil*, Aronia melanocarpa (Chokeberry) seed oil*, Vaccinium macrocarpon (Cranberry) seed oil*, Moringa oleifera (Moringa) seed oil**, Persea americana (Avocado) oil*, Ribes nigrum (Black currant) seed oil*, Copaifera officinalis (Copaiba) resin*, Canabis sativa (Hemp) seed oil*, Moringa peregrina seed oil extract & Caprylic/Capric Triglyceride** (Moringa peregrina extract), Ascorbyl tetraisopalmitate (Vitamin C), Proprietary full-spectrum blend of Cannabis sativa (Hemp) extract, Silica (Algica), Ergocalciferol (Vitamin D2), Menaquinone (Vitamin K2), Tocopherol (Vitamin E)* Organic Ingredient* Wild Crafted/Regenerative**
  Other Names: Hemptress Multifunction Oil

SUMMARY:
For the skin to function optimally, it needs to be nourished and supplied with the necessary compounds to support health. However, many individuals are deficient in those compounds, leading to negative skin outcomes. Most products on the market today only supply one or two compounds that can benefit skin health. Hemptress has developed a multi-function oil designed to help with outcomes related to acne, aging, and eczema, among others.

This twelve-week trial will examine the effectiveness of Hemptress' test product. This study will be a two-group trial with 45 participants per group. One group will focus on understanding the test product's effects on skin aging symptoms. The other group will focus on understanding the test product's effects on acne and eczema. The trial will be hybrid, and the participants will follow the use instructions provided by the research team.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in the Acne and Eczema group in this study, an individual must meet all of the following criteria:

* Male or Female between 21-55 years of age.
* Must be in good general health.
* Must experience regular acne, pimples, eczema, or blemishes.
* Must be willing to maintain the following skincare routine during the study: (1)Daily cleansing or rinsing of their face in the morning or the evening is sufficient. We prefer less daily cleansing vs. more. If males go in the shower and rinse, that is sufficient. (2) The option to wear sunscreen if the sunscreen brand is pre-approved - a person who does not wear sunscreen is more desirable. The test product does contain some sun protection (3) - Must NOT use any moisturizer besides our oil. Must use the test product in the morning and the evening daily. Must not be using retinoids and must not start using retinoids during the study. Must NOT use oral anti-acne medications/prescriptions.
* Must not be using retinoids.
* Must be willing to comply with the protocol.

To be eligible to participate in the Anti-Aging group in this study, an individual must meet all of the following criteria:

* Male or Female between 40-65 years of age
* Must be in good general health.
* Must experience early-stage wrinkles not treated by topical or oral prescription drugs/medication or over-the-counter products
* May experience hyperpigmentation and dark spots.
* Must be willing to maintain the following skincare routine during the study: (1)Daily cleansing or rinsing their face in the morning or the evening is sufficient. We prefer less daily cleansing vs. more. If males just go in the shower and rinse, that is fine. (2) The option to wear sunscreen if the sunscreen brand is pre-approved - a person who does not wear sunscreen is more desirable. The test product does contain some sun protection. (3) - Must NOT use any moisturizer besides our oil. Must be willing to use the test product in the morning and the evening.
* Must not be using retinoids.
* Must be willing to comply with the protocol.
* Is willing to come to the Citruslabs office for pictures of their skin to be taken at baseline and at the end of the study.

Exclusion Criteria:

An individual who meets the following criteria will be excluded from participation in this study in the Acne and Eczema Group:

* Females who are pregnant or breastfeeding
* Unwilling to follow the protocol.
* Unwilling to discontinue using all moisturizers except for the test product during the trial.
* Currently participating in another study.
* Usage of an oral acne treatment
* Use of a prescription medication relevant to the skin.
* Anyone undergoing cosmetic procedures during the study, including Botox, laser, or chemical peel treatments.
* Anyone sensitive or allergic to any ingredients found in the products.
* Anyone with learning or cognitive difficulties that would prevent them from reading and understanding questionnaires and surveys.
* Anyone with severe chronic conditions, including oncological conditions, psychiatric disorders or diabetes.
* Anyone who uses sunscreen that is mineral-based can participate if the brand is pre-approved.

An individual who meets the following criteria will be excluded from participation in this study in the Anti-Aging Group:

* Females who are pregnant or breastfeeding
* Unwilling to follow the protocol.
* Unwilling to discontinue using all moisturizers except for the test product during the trial.
* Currently participating in another study.
* Usage of products that include chemical exfoliating ingredients such as glycolic acid, lactic acid, or salicylic acid.
* Use of oral or topical retinoids
* Individuals with cystic acne or otherwise very acne-prone skin.
* Individuals experiencing strong bouts of hormonal acne.
* Use of a prescription medication relevant to the skin.
* Anyone undergoing cosmetic procedures during the study, including Botox, laser, or chemical peel treatments.
* Anyone sensitive or allergic to any ingredients found in the products.
* Anyone with learning or cognitive difficulties that would prevent them from reading and understanding questionnaires and surveys.
* Anyone with severe chronic conditions, including oncological conditions, psychiatric disorders or diabetes.
* Anyone who uses sunscreen that is mineral-based can participate if the brand is pre-approved.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Skin Health [Time Frame: Baseline to Week 12] | 12 weeks
  Survey-based assessment of participant-perceived changes in skin health. Assessed using 0-5 point Likert scale, with 0 representing the most beneficial outcome (no symptoms) and 5 representing the worst outcome (severe symptoms).

SECONDARY OUTCOMES:
Change in VISIA® Skin Analysis Score [Time Frame: Baseline to Week 12] | 12 weeks
  VISIA® Skin Analysis system will be used to assess changes in skin outcomes. Analysis will be conducted by a board-certified dermatologist at Baseline and Week 8. The VISIA® Skin Analysis system will be used to capture the images which will then be processed by the VISIA software. The software utilizes advanced algorithms to detect and measure specific skin attributes. The skin attributes/parameters evaluated will be Wrinkles, Spots, Pores, Texture, Redness and UV Damage. These parameters are evaluated using the captured images and the specialized algorithms employed by the VISIA software. The results are then used to generate a comprehensive analysis report, which includes both the quantitative measurements and qualitative assessments, along with any corresponding scores or ratings assigned to different skin attributes. Mean participant's scores for each parameter will be calculated at Baseline and Week 8 and compared for statistical significance.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States